CLINICAL TRIAL: NCT06425536
Title: Efficacy of Remineralizing Products Used in Molar Grooves: RCT With Evaluation With Diagnodent Pen and Diagnocam
Brief Title: Efficacy of Remineralizing Products Used in Molar Grooves: Evaluation With Diagnodent Pen and Diagnocam
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pavia (Other)
Responsible Party: Principal Investigator, Andrea Scribante, Associate Professor, Principal Investigator, University of Pavia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2024-MOLARGROOVES
Record Dates: First submitted 2024-05-17; First posted 2024-05-22 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Enamel Caries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biorepair Total protection toothpaste (Experimental)
  Interventions: Other: Home use
- Biosmalto Caries and Erosion (Active Comparator)
  Interventions: Other: Home use

INTERVENTIONS:
Other: Home use — Home use twice a day

SUMMARY:
To evaluate the efficacy of enamel remineralization by biomimetic hydroxyapatite contained in microRepair-based Biorepair Total Protection toothpaste compared to the use of Bio Enamel Caries and Erosion toothpaste based on Fluoro-Hydroxyapatite and BioActive Complex, evaluated with Diagnodent Pen and Diagnocam.

DETAILED DESCRIPTION:
The recruited patients will be divided into:

Group 1: Active group 20 patients undergoing quarterly oral hygiene sessions and home treatment using Biorepair Total Protection toothpaste 2 times/day

Gruppo 2: Active group 20 patients undergoing quarterly oral hygiene sessions and home treatment using Curasept Biosmalto Caries and Erosion toothpaste 2 times/day

For both groups, Diagnodent Pen will be used to evaluate the degree of demineralization, while Diagnocam will be used as qualitative evaluation.

Other clinical indices to be collected are: plaque index (PI), bleeding index (BOP), basic erosive wear examination (BEWE), Schiff Air Index (SAI).

The time frames of the study are:

* T0: baseline
* T1: after 1 month
* T2: after 3 months
* T3: after 6 months

ELIGIBILITY:
Inclusion Criteria:

* First permanent molars erupted and completely healthy
* Patients presenting C1 values 0-12 and C2 values 13-24 of the Diagnodent Pen

Exclusion Criteria:

* Patients with Diagnodent-stimulated value > 25
* Patients with groove sealings of sealed permanent first molars or composite restorations
* First molars with extensive demineralizations (Molar Incisor Hypomineralization, fluorosis, white/brown spots)

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-11-25 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Change in Diagnodent Pen value | Study begin, 1, 3 and 6 months after the baseline
  Scores (according to the manufacturer):
  0 - 12: Normal prophylaxis (such as fluoride toothpaste) 13 - 24: Intensive prophylaxis (e.g. fluoridation, remineralisation) > 25: Minimally invasive restorative procedures, composite filling materials and intensive prophylaxis (e.g. remineralisation, Air Abrasion, SONICflex micro), conventional restoration with large lesions, depending on risk assessment and findings.
Change in Diagnocam value | Study begin, 1, 3 and 6 months after the baseline
  Qualitative evaluation.
Change in Schiff Air Index | Study begin, 1, 3 and 6 months after the baseline
  0: the subject did not respond to air blasting;
  1. the subject responded to air blasting;
  2. the subject responded to air blasting and requested discontinuation;
  3. the subject responded to air blasting, requested discontinuation and considered the stimulus to be painful.
Change in Bleeding on Probing | Study begin, 1, 3 and 6 months after the baseline
  Site-specific assessment of the presence or absence of gum bleeding after the insertion of the periodontal probe for the detection of PPD, detected on 6 sites.
  Percentage of sites with bleeding on probing determines the BOP%.
Change in Plaque Index | Study begin, 1, 3 and 6 months after the baseline
  Evaluation of the presence of plaque on the 4 surfaces of teeth on the total amount of dental surfaces.
  Formula = n ° sites with plaque / total n ° of dental surfaces x100
Change in Basic Erosive Wear Examination | Study begin, 1, 3 and 6 months after the baseline
  Scoring criteria (Barlet et al., 2008):
  0: no erosive tooth wear;
  1. initial loss of surface texture;
  2. distinct defect, hard tissue loss < 50% of the surface area;
  3. hard tissue loss ≥ 50% of the surface area.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Scribante, DDS, PhD, Principal Investigator — University of Pavia
Locations (1):
- Unit of Dental Hygiene - Section of Dentistry - Department of Clinical, Surgical, Diagnostic and Paediatrics - University of Pavia, Pavia, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No
Data will be available upon motivated request to the Principal Investigator.